CLINICAL TRIAL: NCT05028088
Title: Diaphragm Ultrasound to Evaluate the Antagonistic Effect of Sugammadex on Rocuronium After Liver Surgery in Patients With Different Liver Child-Pugh Grades
Brief Title: Diaphragm Ultrasound to Evaluate the Antagonistic Effect of Sugammadex
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2016Summer
Record Dates: First submitted 2021-07-18; First posted 2021-08-31 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Diaphragm Ultrasonography; Liver Dysfunction; Sugammadex; Rocuronium
MeSH Terms: conditions — Liver Diseases | interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Child-Pugh A (Experimental): 1. Diaphragm ultrasound scan before induction of anesthesia.
  2. Anesthesia method: During anesthesia induction, propofol 2.5mg/kg and sufentanil 5μg/kg will be injected intravenously. When the BIS value drops below 60, the muscle relaxation monitor will be calibrated. After T1 and TOF are stable, rocuronium will be injected intravenously at 0.6 mg/kg. During the maintenance stage of anesthesia, the pneumoperitoneum pressure will be at a low level of 8-10mmHg, propofol TCI will be applied to maintain the plasma concentration of 2.5-5.5 μg/mL, remifentanil TCI will be used to keep the plasma concentration of 0.5-5 ng/mL, and rocuronium will be continuously pumped intravenously with 0.3-0.6 mg/kg/h for deep muscle relaxations, with the the post-tetanic twitch count (PTC) value of 1 to 2.
  3. When the TOF value was ≥2%, patients in each group will be given SUG (2mg/kg).
  4. Diaphragm ultrasound scan at the immediate time,10min, 30min and 2h after extubation.
  Interventions: Drug: sugammadex
- Child-Pugh B (Experimental): 1. Diaphragm ultrasound scan before induction of anesthesia.
  2. Anesthesia method: During anesthesia induction, propofol 2.5mg/kg and sufentanil 5μg/kg will be injected intravenously. When the BIS value drops below 60, the muscle relaxation monitor will be calibrated. After T1 and TOF are stable, rocuronium will be injected intravenously at 0.6 mg/kg. During the maintenance stage of anesthesia, the pneumoperitoneum pressure will be at a low level of 8-10mmHg, propofol TCI will be applied to maintain the plasma concentration of 2.5-5.5 μg/mL, remifentanil TCI will be used to keep the plasma concentration of 0.5-5 ng/mL, and rocuronium will be continuously pumped intravenously with 0.3-0.6 mg/kg/h for deep muscle relaxations, with the the post-tetanic twitch count (PTC) value of 1 to 2.
  3. When the TOF value was ≥2%, patients in each group will be given SUG (2mg/kg).
  4. Diaphragm ultrasound scan at the immediate time,10min, 30min and 2h after extubation.
  Interventions: Drug: sugammadex
- Child-Pugh C (Experimental): 1. Diaphragm ultrasound scan before induction of anesthesia.
  2. Anesthesia method: During anesthesia induction, propofol 2.5mg/kg and sufentanil 5μg/kg will be injected intravenously. When the BIS value drops below 60, the muscle relaxation monitor will be calibrated. After T1 and TOF are stable, rocuronium will be injected intravenously at 0.6 mg/kg. During the maintenance stage of anesthesia, the pneumoperitoneum pressure will be at a low level of 8-10mmHg, propofol TCI will be applied to maintain the plasma concentration of 2.5-5.5 μg/mL, remifentanil TCI will be used to keep the plasma concentration of 0.5-5 ng/mL, and rocuronium will be continuously pumped intravenously with 0.3-0.6 mg/kg/h for deep muscle relaxations, with the the post-tetanic twitch count (PTC) value of 1 to 2.
  3. When the TOF value was ≥2%, patients in each group will be given SUG (2mg/kg).
  4. Diaphragm ultrasound scan at the immediate time,10min, 30min and 2h after extubation.
  Interventions: Drug: sugammadex

INTERVENTIONS:
Drug: sugammadex — This study is a prospective, double-blind, low-intervention, non-randomized controlled clinical trial involving 99 patients with American Society of Anesthesiologists Ⅰ-Ⅲ, body mass index 18.5-24.9 kg/m2, who will undergo laparoscopic radical resection of liver cancer under general anesthesia in the Wuhan Union Hospital. Ultrasonography will be applied to monitor the change rate of diaphragm thickness at different time after extubation to evaluate the recovery rate of muscle relaxant, which indirectly reflects the dose-effect relationship of SUG antagonizing against rocuronium in patients with different liver Child-Pugh grades preoperatively.
  Other Names: diaphragm ultrasonography

SUMMARY:
The use of muscle relaxants is an indispensable in the general anesthesia but is prone to accidents, which are often related to residual muscle relaxant. Therefore, how to timely and effectively eliminate the residual effect of muscle relaxants after surgery has become an urgent clinical problem. Rocuronium is a non-depolarizing muscle relaxant that is primarily metabolized by the liver. Patients with liver dysfunction can affect the metabolic process of rocuronium, thereby delaying the recovery of muscle relaxation. Sugammadex (SUG) is a novel specific antagonist of aminosteroid muscle relaxants, which can effectively antagonize muscle relaxants at different depths. However, whether liver dysfunction affects the antagonistic effect of SUG against rocuronium has not been reported yet. Therefore, the investigators hypothesize that with the increase of patients' liver Child-Pugh grade, the recovery time of rocuronium antagonized by the same dose of SUG after surgery will be prolonged, and the incidence of muscle relaxation residual will be increased in the short term.

DETAILED DESCRIPTION:
Main instruments: Drager Fabius anesthesia machine, interlive vue MX600 monitor, Train-Of-Four-Watch muscle relaxation monitor, Philips IU22 Color Doppler Ultrasound Diagnostic Instrument.

Diaphragm ultrasound scan: Prior to anesthesia induction, patients will lie on the bed in a semi-recumbent (45°) position. One operator skilled in ultrasonography will identify and locate diaphragm using the hyperechoic pleural and peritoneal layers with an Philips IU22 Color Doppler Ultrasound Diagnostic Instrument.

Anesthesia method: After the patient entered the operating room, venous access will be opened in the forearm, and routine monitoring of non-invasive BP, ECG, oxygen saturation(SpO₂) and bispectral index(BIS) will be performed. During anesthesia induction, propofol 2.5mg/kg and sufentanil 5μg/kg will be injected intravenously. When the BIS value drops below 60, the muscle relaxation monitor will be calibrated. After T1 and TOF are stable, rocuronium will be injected intravenously at 0.6 mg/kg. By the time T1=0, endotracheal intubation will be given, and the respiratory parameters will need to be adjusted to volume control ventilation (VT 8-10 ml/kg, respiratory rate(RR) 12-18 times/min, and PETCO2 35-45 mmHg). During the maintenance stage of anesthesia, the pneumoperitoneum pressure will be at a low level of 8-10mmHg, propofol target-controlled infusion(TCI) will be applied to maintain the plasma concentration of 2.5-5.5 μg/mL, remifentanil TCI will be used to keep the plasma concentration of 0.5-5 ng/mL, and rocuronium will be continuously pumped intravenously with 0.3-0.6 mg/kg/h for deep muscle relaxations, with the the post-tetanic twitch count (PTC) value of 1 to 2.

Muscle relaxation monitoring: TOF-Watch SX muscle relaxation monitor is going to be adopted in our study. The investigators will standardize the electrode position of the muscle relaxation monitor. The distal electrode will be placed at the intersection of the radial edge of the ulnar flexor carpi and the proximal edge of the wrist curve, while the proximal electrode will be placed 3-6 cm away from the distal electrode. Two electrodes will put on either side of the predicted location of the ulnar nerve, which will be able to minimize the impact caused by misjudgment of the location of the nerve.

Measurement of diaphragmatic thickness: When B-mode ultrasound will be used to measure the thickness of the diaphragm, a 5-12MHz linear array ultrasound probe will be put in the left midaxillary line between the 8-10 costale, where is called the diaphragmatic zone of apposition (ZAP). In the breathing exercise, the diaphragm is relatively fixed at ZAP, and the breathing action has little influence on the movement of the diaphragm at ZAP, the diaphragm only shows systolic and diastolic changes. Therefore, the measurement of the diaphragm thickness at ZAP can truly reflect the overall thickness change of the diaphragm during the respiratory cycle. Each value will be measured three times in three consecutive breathing cycles, and the average of the nine measurements will be taken. The values of diaphragmatic thickness at the end of inspirations (DTEI) and diaphragmatic thickness at the end of expirations (DTEE) will be recorded respectively, then the change rate of diaphragmatic thickness fraction (DTF) = (DTEI - DTEE) / DTEE × 100% will be calculated. In addition, the recover rate of DTF = (pre-anesthetic DTEI - postoperative DTEI) / pre-anesthetic DTEI × 100% also will be figured out. Ultrasound measurements should be performed by two physicians with ultrasound experience. Results will be kept confidential to the investigator, who will analyze the ultrasound data when the research is over.

The infusion of anesthetic drugs should be stopped at the end of surgery, and the patients will be transferred into the Post-Anesthesia Care Unit (PACU) with endotracheal catheters and continued monitoring. When the TOF value was ≥2%, patients in each group will be given SUG (2mg/kg), respectively. The researchers will record the recovery conditions of diaphragmatic function monitored by bedside ultrasound at the immediate time,10min, 30min and 2h after extubation.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age between 18 and 65 years old.
* 2.Patients scheduled for laparoscopic radical resection of liver cancer under general anesthesia.
* 3.Patients ASA classification Ⅰ-Ⅲ.
* 4.Body mass index 18.5 kg/m2 ~ 24.9 kg/m2
* 5.Able to give informed consent.
* 6.The surgical position is suitable for BIS monitoring and muscle relaxation monitoring.

Exclusion Criteria:

* 1.Patients with allergic to rocuronium and SUG.
* 2.Patients with central and peripheral nervous system diseases, such as polio, Parkinson's disease, peripheral neuropathy, etc..
* 3.Patients with neuromuscular system diseases, such as multiple sclerosis, myasthenia gravis, atrophic myotonia, etc..
* 4.Patients with diaphragm dysfunction, pneumothorax, pleural effusion, mediastinal pneumatosis.
* 5.Pregnant women or nursing mothers.
* 6.Judging by the researchers, patients with other conditions who are unsuitable for clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
the recovery rate of muscle relaxation | 2 hours
  the incidence of residual muscle relaxation at different time points after the operation and the baseline recovery rate of the diaphragm（immediately after extubation, 10minutes, 30minutes and 2hours）
  When the patients' consciousness and spontaneous breathing are restored, participants can open their eyes according to the doctor's instructions, shake hands firmly, and at the same time, participants can complete the movement of raising their head continuously for more than 5 seconds to remove the tracheal tube.

SECONDARY OUTCOMES:
muscle relaxation onset time | within 3 minutes
  the period from administration of rocuronium to tracheal intubation
intraoperative rocuronium dosage | through anesthesia completion, up to 2 hours
  The sum of the dose of rocuronium bromide used in induction and maintenance of anesthesia.
PACU monitoring time | about 2 hours
  Total time patients are monitored in PACU after surgery.
the incidence of postoperative pulmonary complications | within 7 days after surgery
  incidence of postoperative pulmonary complications within seven days

CONTACTS AND LOCATIONS:
Overall Officials: Yun Lin, MD, PhD., Principal Investigator — Union Hospital of Tongji Medical College of Huazhong University of Science and Technology
Locations (1):
- Union Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
The investigators don not plan to make the IPD collected in this study available to other researchers.

REFERENCES:
- [Background] Whittaker R, Wedell D. Review of neuromuscular blockers. Compendium. 1991 Jun;12(6):408, 410, 412 passim. PMID 1718602
- [Background] Naguib M, Magboul MM. Adverse effects of neuromuscular blockers and their antagonists. Drug Saf. 1998 Feb;18(2):99-116. doi: 10.2165/00002018-199818020-00002. PMID 9512917
- [Background] Arino-Irujo JJ, Calbet-Manueco A, De la Calle-Elguezabal PA, Velasco-Barrio JM, Lopez-Timoneda F, Ortiz-Gomez JR, Fabregat-Lopez J, Palacio-Abizanda FJ, Fornet-Ruiz I, Perez-Cajaraville J. [Neuromuscular blockade monitoring. Part 1]. Rev Esp Anestesiol Reanim. 2010 Mar;57(3):153-60. doi: 10.1016/s0034-9356(10)70190-0. Spanish. PMID 20422848
- [Background] Fuchs-Buder T, Schmartz D. [Residual neuromuscular blockade]. Anaesthesist. 2017 Jun;66(6):465-476. doi: 10.1007/s00101-017-0325-1. German. PMID 28573344
- [Background] Brull SJ, Kopman AF. Current Status of Neuromuscular Reversal and Monitoring: Challenges and Opportunities. Anesthesiology. 2017 Jan;126(1):173-190. doi: 10.1097/ALN.0000000000001409. PMID 27820709
- [Background] Murphy GS, Brull SJ. Residual neuromuscular block: lessons unlearned. Part I: definitions, incidence, and adverse physiologic effects of residual neuromuscular block. Anesth Analg. 2010 Jul;111(1):120-8. doi: 10.1213/ANE.0b013e3181da832d. Epub 2010 May 4. PMID 20442260
- [Background] Aytac I, Postaci A, Aytac B, Sacan O, Alay GH, Celik B, Kahveci K, Dikmen B. Survey of postoperative residual curarization, acute respiratory events and approach of anesthesiologists. Braz J Anesthesiol. 2016 Jan-Feb;66(1):55-62. doi: 10.1016/j.bjane.2012.06.011. Epub 2014 Apr 4. PMID 26768931
- [Background] Shay D, Wongtangman K, Eikermann M, Schaefer MS. The effects of acetylcholinesterase inhibitors on morbidity after general anesthesia and surgery. Neuropharmacology. 2020 Aug 15;173:108134. doi: 10.1016/j.neuropharm.2020.108134. Epub 2020 May 19. PMID 32416089
- [Background] Hawkins J, Khanna S, Argalious M. Sugammadex for Reversal of Neuromuscular Blockade: Uses and Limitations. Curr Pharm Des. 2019;25(19):2140-2148. doi: 10.2174/1381612825666190704101145. PMID 31272347
- [Background] Tao J, Zhang W, Yue H, Zhu G, Wu W, Gong W, Fang H, He G, Hu X, Zhao H, Liu A. Prevalence of Hepatitis B Virus Infection in Shenzhen, China, 2015-2018. Sci Rep. 2019 Sep 26;9(1):13948. doi: 10.1038/s41598-019-50173-5. PMID 31558731
- [Derived] Sun Y, Sun S, Chen R, Shen J, Chen X, Lin Y, Yao S. Diaphragm ultrasonography as a monitor in assessing antagonistic effect of sugammadex on rocuronium in patients with Child-Pugh grades A and B. Front Med (Lausanne). 2024 Apr 5;11:1370021. doi: 10.3389/fmed.2024.1370021. eCollection 2024. PMID 38686365
- [Derived] Sun S, Sun Y, Chen R, Yao C, Xia H, Chen X, Lin Y, Yao S. Diaphragm ultrasound to evaluate the antagonistic effect of sugammadex on rocuronium after liver surgery in patients with different liver Child-Pugh grades: study protocol for a prospective, double-blind, non-randomised controlled trial. BMJ Open. 2022 Feb 1;12(2):e052279. doi: 10.1136/bmjopen-2021-052279. PMID 35105573